CLINICAL TRIAL: NCT07305376
Title: Older Adults' Attitudes Towards Stopping Aspirin
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Sarah Vordenberg, Associate Chair and Clinical Professor Department of Clinical Pharmacy, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00280646
Record Dates: First submitted 2025-11-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Medication Overuse
MeSH Terms: conditions — Prescription Drug Overuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Source of recommendation - Physician (Experimental): Participants read a hypothetical scenario where a doctor recommends stopping aspirin.
  Interventions: Other: Additional harm information; Other: Less information
- Source of recommendation - Pharmacist (Experimental): Participants read a hypothetical scenario where a pharmacist recommends stopping aspirin.
  Interventions: Other: Additional harm information; Other: Less information
- Source of information - AI (Experimental): Participants read a hypothetical scenario where artificial intelligence is used to recommend stopping aspirin.
  Interventions: Other: Additional harm information; Other: Less information

INTERVENTIONS:
Other: Additional harm information — Participants received additional information about the harm of continuing aspirin.
Other: Less information — Participants will receive less information about the risk of harms of continuing aspirin.

SUMMARY:
This online, survey-based experiment will include 2,400 adults who are 65 years and older (n=1,200 each from the United States and Australia). Each participant will be asked to share their opinions on a hypothetical patient scenario developed by our multidisciplinary team. This work is expected to significantly contribute to the understanding of how older adults make decisions about deprescribing medications. The long-term goal is to enhance communication between older adults and clinicians so that medication regimens are optimized and align with care preferences. These results will directly inform future research on the impact of communication choices in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Australia or the United States
* 65 years and older

Exclusion Criteria:

* Unable to read survey written in English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
"How safe do you think it would be to continue taking aspirin?" measured on a 6-point Likert scale | Day 1
"How helpful do you think it would be to continue taking aspirin?" measured on a 6-point Likert scale | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Vordenberg, PharmD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No